CLINICAL TRIAL: NCT06821724
Title: Comparative Study on the Effect of Different Remineralizing Agents Versus Fluoride Gel on White Spot Lesions After In-Office Followed by Home Treatment in Children: A Randomized Controlled Clinical Study
Brief Title: Effect of Different Remineralizing Agents on White Spot Lesions Treatment in Children
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Mohamed Farouk Rashed, Researcher of Pediatric Dentistry, National Research Centre, Egypt
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 342
Record Dates: First submitted 2025-02-06; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: White Spot Lesion of Tooth
Keywords: White spots; Remineralization; Caries; Children
MeSH Terms: interventions — casein phosphopeptide-amorphous calcium phosphate nanocomplex; Fluorides

STUDY DESIGN:
Intervention Model Description: Randomized controlled parallel double blinded study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Blinding to the child participants and legal guardian of each participating child, inter examiner and statistician. The operator and the child were blinded to the intervention from the beginning till teeth polishing. Blinding cannot be done during application of remineralizing agents because of clear visual differences between these agents.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- No treatment (No Intervention): Negative control
- Fluoride gel (Active Comparator): Positive control
  Interventions: Drug: Fluoride gel
- Casein phosphopeptide-amorphous calcium phosphate (CPP-ACP) (MI paste) (Experimental): Intervention
  Interventions: Drug: Casein phosphopeptide-amorphous calcium phosphate
- Casein phosphopeptide-amorphous calcium phosphate (CPP-ACP) + fluoride (MI paste plus) (Experimental): Intervention
  Interventions: Drug: Casein phosphopeptide-amorphous calcium phosphate + fluoride
- Nano hydroxyapatite paste (Apagard primo toothpaste) (Experimental): Intervention
  Interventions: Drug: Nano hydroxyapatite paste

INTERVENTIONS:
Drug: Casein phosphopeptide-amorphous calcium phosphate — Intervention
  Other Names: (CPP-ACP) (MI paste)
  Arms: Casein phosphopeptide-amorphous calcium phosphate (CPP-ACP) (MI paste)
Drug: Casein phosphopeptide-amorphous calcium phosphate + fluoride — Intervention
  Other Names: (CPP-ACP) + (MI paste plus)
  Arms: Casein phosphopeptide-amorphous calcium phosphate (CPP-ACP) + fluoride (MI paste plus)
Drug: Nano hydroxyapatite paste — Intervention
  Other Names: (Apagard primo toothpaste)
  Arms: Nano hydroxyapatite paste (Apagard primo toothpaste)
Drug: Fluoride gel — Positive control
  Other Names: Active Comparator
  Arms: Fluoride gel

SUMMARY:
One hundred children with white spot lesions on their teeth were divivided into 5 groups of different remineralizing agents to assess their effect on color change and remineralization

DETAILED DESCRIPTION:
Children having at least one tooth clinically diagnosed by white spot lesion were randomly allocated to five groups.

Group one: No treatment was applied (negative control). Group two: Fluoride gel was applied for 5 minutes (positive control). Group three: Casein phosphopeptide-amorphous calcium phosphate (CPP-ACP) (MI paste) was applied for 5 minutes.

Group four: Casein phosphopeptide-amorphous calcium phosphate (CPP-ACP) + fluoride (MI paste plus) were applied for 5 minutes.

Group five: Nano hydroxyapatite paste (Apagard primo toothpaste) was be applied for 5 minutes.

All children involved in this study were instructed to brush their teeth under the supervision of the researcher before the application of the studied agent.

Each agent was applied to the labial surfaces of each tooth affected with white spot lesion for 5 minutes after cleaning and drying with a cotton roll using an applicator tip. After each application, children were instructed not to eat or drink for one hour. This application was be repeated in-office after one then after two weeks then after six weeks.

Participants received a sterilized pouch containing a sterile container with one of the pastes according to the study group for home application. The application of the paste was carried out under parental supervision and was asked to apply each of the pastes at home three times a day till the end of the study

ELIGIBILITY:
Inclusion Criteria:

1. Presence of at least one tooth affected by white spot lesion.
2. Good oral hygiene and regular tooth brushing at least twice daily.

Exclusion Criteria:

1. Unwillingness to be randomly assigned to 1 of the 3 treatment groups.
2. Presence of abnormal oral, medical, or mental condition.
3. Presence of any milk-related allergies.
4. Presence of dentin caries or enamel hypoplasia on maxillary anterior teeth.
5. Presence of periodontal pockets around maxillary anterior teeth.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Assessment of color change | before treatment, immediately after treatment, 2 weeks and 6 weeks after the onset of treatment
  Color change assessmentof white spot lesions using "Easy-shade" device

SECONDARY OUTCOMES:
Remineralization assessment | before treatment, immediately after treatment, 2 weeks and 6 weeks after the onset of treatment
  Remineralization assessment will be done using Laser fluorescence device "DIAGNOdent® (KaVo)".

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed F Rashed, Researcher, Study Director — National Research Centre, Egypt
Locations (1):
- National Research Centre, Dokki, Giza Governorate, Egypt

REFERENCES:
- [Derived] El Mansy MM, Rashed MF, Saleh RS. Effect of remineralization after in office followed by home treatment of white spot lesions in children randomized controlled trial. Sci Rep. 2025 Aug 19;15(1):30448. doi: 10.1038/s41598-025-15829-5. PMID 40830200